CLINICAL TRIAL: NCT02863185
Title: Effect of Pitavastatin on Erythrocyte Membrane Fatty Acid Contents in Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, WON SUK AN, Professor, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pita_2016
Record Dates: First submitted 2016-08-01; First posted 2016-08-11 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; pitavastatin; erythrocyte membrane fatty acid
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — pitavastatin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pitavastatin group (Experimental): Use of 2mg or 4mg Pitavastatin
  Interventions: Drug: Pitavastatin
- Atorvastatin group (Active Comparator): Use of 10mg or 20mg Atorvastatin
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Pitavastatin
  Arms: Pitavastatin group
Drug: Atorvastatin
  Arms: Atorvastatin group

SUMMARY:
Patients with chronic kidney disease (CKD) are high risk for death and cardiac disease is the major cause of death. CKD patients commonly have traditional risk factors for coronary artery disease, such as age, gender, hypertension, cigarette smoking, and dyslipidemia. Previous studies have reported that reducing cholesterol levels is associated with reducing morbidity and mortality from atherosclerosis. In particular, pharmacologic treatment using statin has been decreased the risk of adverse cardiovascular events in CKD population. Therefore, guidelines recommended the use of statin in CKD patients. On the other hands, niacin or fibrates is not recommended concomitantly with statins in patients with CKD because of increased risk of adverse events. In addition, recent study has reported that there was no incremental clinical benefit from the addition of niacin to statin therapy, in further decreasing the incidence of major cardiac events.

Supplementation with omega-3 fatty acid (FA) lowers the risk of cardiovascular death in patients with myocardial infarction. This cardioprotective effect of omega-3 FA can be explained by anti-inflammatory, anti-oxidative, or anti-thrombic effects. In addition, omega-3 FA modulates cell membrane receptors and affects signal transduction and eicosanoid metabolism. The erythrocyte membrane content of FA has been shown to correlated with the FA content of the myocardium. The risk of cardiovascular disease is significantly reduced in patients with high omega-3 FA, such as eicosapentanoic acid or docosahexaenoic acid (DHA), in the erythrocyte membrane. In contrast, high levels of erythrocyte membrane total trans-FA, trans-oleic acid, and arachidonic acid (AA) are associated with an increased risk of cardiovascular disease. Erythrocyte membrane monounsaturated FA (MUFA) content, including oleic acid, is significantly higher in patients with acute coronary syndrome than control subjects. The erythrocyte membrane oleic acid content was also higher in dialysis patients who have high risks of cardiovascular disease compared to control subjects. Therefore, the modification of erythrocyte membrane FA content is very important with respect to cardiovascular disease. In a previous study, erythrocyte membrane omega-3 FA was shown to be increased and the MUFA content was decreased after omega-3 FA supplementation in HD patients. However, there are no reports about the effect of statin on the erythrocyte membrane FA composition in CKD. Recent study has reported that those with pitavastatin 4mg were decreased DHA to AA ratio, but those with pravastatin 20 mg were not change the DHA to AA ratio in patient with CAD. Statin may have important role on the modulation of erythrocyte membrane FA. In this study, the investigators hypothesized that pitavastatin supplementation can modify erythrocyte membrane FA content, including MUFA and oleic acid, in CKD patients. In addition, the investigators evaluated the effect of pitavastatin on adiponectin and glucose level in CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients who agreed with written informed consent
* CKD patients who do not taking statin agent.
* Who have LDL cholesterol over 100mg/dL and coronary vascular disease(CVD) or equivalent risk; Who have LDL cholesterol over 130mg/dL and two or more coronary vascular risk; Whose LDL cholesterol over 160mg/dL in patient with CKD stage 1 to 5 without dialysis.

Exclusion Criteria:

* Patients with acute illness, a history of active infection, CVD, acute kidney injury during the past 3 months, or a history of malignancy or liver disease
* Patients using statin, omega-3 fatty acid or sevelamer hydrochloride within 3 months
* Patients who experienced side effects by statin treatment
* Pregnant or pregnancy expected CKD patients
* Patient with dyslipidemia due to nephrotic syndrome
* Patient taken imaging study using contrast media during the past 14 days
* Patient with albumin level < 3.0 g/dL

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
mean difference and change of erythrocyte membrane fatty acid including oleic acid | baseline and 24 weeks after intervention

SECONDARY OUTCOMES:
mean difference and change of total cholesterol, triglyceride, LDL-cholesterol, HDL-cholesterol | baseline and 24 weeks after intervention
mean difference and change of adiponectin | baseline and 24 weeks after intervention
mean difference and change of glucose and glycosylated hemoglobin | baseline and 24 weeks after intervention
mean difference and change of proteinuria | baseline and 24 weeks after intervention

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Won Suk An, Busan
  - Dong-A University, Busan

REFERENCES:
- [Background] Tonelli M, Muntner P, Lloyd A, Manns B, Klarenbach S, Pannu N, James M, Hemmelgarn B; Alberta Kidney Disease Network. Association between LDL-C and risk of myocardial infarction in CKD. J Am Soc Nephrol. 2013 May;24(6):979-86. doi: 10.1681/ASN.2012080870. Epub 2013 May 16. PMID 23687359
- [Background] Baigent C, Landray MJ, Reith C, Emberson J, Wheeler DC, Tomson C, Wanner C, Krane V, Cass A, Craig J, Neal B, Jiang L, Hooi LS, Levin A, Agodoa L, Gaziano M, Kasiske B, Walker R, Massy ZA, Feldt-Rasmussen B, Krairittichai U, Ophascharoensuk V, Fellstrom B, Holdaas H, Tesar V, Wiecek A, Grobbee D, de Zeeuw D, Gronhagen-Riska C, Dasgupta T, Lewis D, Herrington W, Mafham M, Majoni W, Wallendszus K, Grimm R, Pedersen T, Tobert J, Armitage J, Baxter A, Bray C, Chen Y, Chen Z, Hill M, Knott C, Parish S, Simpson D, Sleight P, Young A, Collins R; SHARP Investigators. The effects of lowering LDL cholesterol with simvastatin plus ezetimibe in patients with chronic kidney disease (Study of Heart and Renal Protection): a randomised placebo-controlled trial. Lancet. 2011 Jun 25;377(9784):2181-92. doi: 10.1016/S0140-6736(11)60739-3. Epub 2011 Jun 12. PMID 21663949
- [Background] Ridker PM, Pradhan A, MacFadyen JG, Libby P, Glynn RJ. Cardiovascular benefits and diabetes risks of statin therapy in primary prevention: an analysis from the JUPITER trial. Lancet. 2012 Aug 11;380(9841):565-71. doi: 10.1016/S0140-6736(12)61190-8. PMID 22883507
- [Background] Leaf A, Kang JX, Xiao YF, Billman GE. Clinical prevention of sudden cardiac death by n-3 polyunsaturated fatty acids and mechanism of prevention of arrhythmias by n-3 fish oils. Circulation. 2003 Jun 3;107(21):2646-52. doi: 10.1161/01.CIR.0000069566.78305.33. No abstract available. PMID 12782616
- [Result] An WS, Kim SE, Kim KH, Lee S, Park Y, Kim HJ, Vaziri ND. Comparison of fatty acid contents of erythrocyte membrane in hemodialysis and peritoneal dialysis patients. J Ren Nutr. 2009 Jul;19(4):267-74. doi: 10.1053/j.jrn.2009.01.027. PMID 19539181
- [Result] An WS, Lee SM, Son YK, Kim SE, Kim KH, Han JY, Bae HR, Rha SH, Park Y. Omega-3 fatty acid supplementation increases 1,25-dihydroxyvitamin D and fetuin-A levels in dialysis patients. Nutr Res. 2012 Jul;32(7):495-502. doi: 10.1016/j.nutres.2012.06.005. Epub 2012 Jul 20. PMID 22901557
- [Result] Nozue T, Yamamoto S, Tohyama S, Fukui K, Umezawa S, Onishi Y, Kunishima T, Sato A, Nozato T, Miyake S, Takeyama Y, Morino Y, Yamauchi T, Muramatsu T, Hibi K, Michishita I. Effects of statins on serum n-3 to n-6 polyunsaturated fatty acid ratios in patients with coronary artery disease. J Cardiovasc Pharmacol Ther. 2013 Jul;18(4):320-6. doi: 10.1177/1074248412473202. Epub 2013 Jan 15. PMID 23324995
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702